CLINICAL TRIAL: NCT06895551
Title: Prospective Multicenter Study on Early Esophageal Cancer Detection: Circulating Tumor DNA Methylation Biomarkers in Liquid Biopsy
Brief Title: Methylation Biomarkers for Pioneering Early Esophageal Cancer Detection
Status: Completed | Type: Observational
Sponsor: Singlera Genomics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EsoMeth
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Cancer
Keywords: ctDNA methylation; early detection
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case group (malignant lesions): Including esophageal cancer and high-grade intraepithelial neoplasia (HGIN).
- Control group (benign lesions): Including low-grade intraepithelial neoplasia (LGIN), submucosal esophageal cancer, benign esophageal lesions, and benign gastric lesions.

SUMMARY:
Esophageal cancer is a highly aggressive malignancy with poor prognosis, ranking as the sixth leading cause of cancer-related deaths worldwide, particularly prevalent in regions such as East Asia and East Africa. This prospective multicenter study aims to develop and validate a blood-based DNA methylation model for the early detection of esophageal cancer and high-grade intraepithelial neoplasia (HGIN). The study will enroll 500 patients with malignant lesions, including esophageal cancer and HGIN, and 500 patients with benign lesions, including low-grade intraepithelial neoplasia (LGIN), submucosal esophageal cancer, benign esophageal lesions, and benign gastric lesions. Through a comprehensive workflow involving methylation marker screening, model construction, training, and validation, we will identify and optimize methylation biomarkers for esophageal cancer detection. The performance of the methylation-based diagnostic model will be rigorously evaluated, including its sensitivity, specificity, and accuracy in distinguishing malignant from benign lesions. This study has the potential to establish a non-invasive, blood-based diagnostic tool for early esophageal cancer detection, which could significantly improve patient outcomes by enabling timely intervention and treatment. The results will contribute to advancing precision medicine in oncology and provide a foundation for future large-scale clinical applications.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, regardless of gender.
2. Willing to undergo gastroscopy or able to provide postoperative esophageal biopsy pathological results.
3. Newly diagnosed esophageal cancer patients (Stage I-IV) who have not undergone surgery, radiotherapy, chemotherapy, targeted therapy, or other tumor-related interventions prior to blood collection (for patients requiring neoadjuvant therapy, blood collection should be performed 1-2 days before neoadjuvant therapy; for patients not requiring neoadjuvant therapy, blood collection should be performed 1-2 days before surgery).

Exclusion Criteria:

1. History of digestive system tumors, including esophageal cancer, gastric cancer, colorectal cancer, liver cancer, etc.
2. History of other cancers that have not achieved clinical cure (clinical cure: no recurrence or metastasis within 5 years post-surgery).
3. Systemic inflammatory response syndrome.
4. Severe cardiovascular disease history (e.g., previous myocardial infarction, coronary artery bypass grafting, or coronary stent implantation; history of congestive heart failure; myocardial infarction within the past 6 months; uncontrolled severe hypertension, etc.) and deemed unsuitable for inclusion by the investigator.
5. Patients who have undergone blood transfusion or major surgical procedures such as transplantation within the past 3 months.
6. Participation in other interventional clinical studies within the past 3 months, or individuals who are pregnant, breastfeeding, or have autoimmune diseases, genetic disorders, mental illnesses, etc.
7. Participation in "interventional" clinical trials and use of investigational drugs within the past 30 days.
8. Other diseases deemed unsuitable for inclusion by the investigator.
9. Failure to adhere to the study plan for timely blood collection.
10. Blood samples that do not meet the requirements (unqualified samples include: ① clotted samples; ② hemolyzed samples; ③ insufficient sample volume; ④ samples delivered for testing more than 72 hours after collection; ⑤ incorrect sample information; ⑥ severe lipemia, with blood appearing milky; ⑦ damaged collection tubes or contaminated samples, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 patients with malignant lesions, including esophageal cancer and HGIN, and 500 patients with benign lesions, including low-grade intraepithelial neoplasia (LGIN), submucosal esophageal cancer, and benign esophageal/gastric lesions
Sampling Method: Non-Probability Sample
Enrollment: 1069 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Methylation Biomarker Panel | assessed up to 36 months
  Evaluate the sensitivity, specificity, and area under the curve (AUC) of the blood-based DNA methylation model in distinguishing esophageal cancer and high-grade intraepithelial neoplasia (HGIN) from benign lesions (including low-grade intraepithelial neoplasia (LGIN), submucosal esophageal cancer, and benign esophageal/gastric lesions).

SECONDARY OUTCOMES:
Model Performance in Subgroups and correlation with Clinical Parameters | assessed up to 36 months
  Assess the diagnostic performance of the methylation model across different subgroups, including early-stage esophageal cancer, advanced-stage esophageal cancer, and HGIN. Investigate the relationship between methylation levels and clinical parameters, including tumor stage (TNM I/II/III/IV), tumor differentiation grade (high/medium/low), age and gender (male/female) etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital, Chinese academy of medical sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No